CLINICAL TRIAL: NCT02416609
Title: Low-dose Radiotherapy as a Chemo-potentiator of a Induction Chemotherapy Regimen With Gem-based Doublets and Stereotactic Body Radiotherapy for Locally Advanced Pancreatic Cancer
Brief Title: Low-dose Radiotherapy Plus Chemotherapy With Gem-based Doublets and Stereotactic Radiotherapy for Advanced Pancreatic Cancer
Acronym: ORCHESTRATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Bruno Meduri, Medical Doctor, Azienda Ospedaliero-Universitaria di Modena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMed1
Record Dates: First submitted 2015-04-07; First posted 2015-04-15 (Estimated); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Pancreatic Cancer
Keywords: Locally advanced pancreatic cancer; Stereotactic Body Radiotherapy; Chemopotentiator; Low dose radiotherapy; Hyper-Radiosensitivity
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gem-based doublets with LDR & sequential SBRT (Experimental): Four Gem-based doublets cycles will be administered concurrent with LDR. If no progression, three fractions of SBRT will be administered.
  Interventions: Radiation: LDR; Drug: Gem-based doublets; Radiation: SBRT

INTERVENTIONS:
Radiation: LDR — LDR will be delivered during each cycle of Gem-based doublets
  Other Names: Low dose radiotherapy
Drug: Gem-based doublets — 4 cycles of Gem-based doublets
Radiation: SBRT — SBRT will be administered after the fourth Gem-based doblet cycle, if no progression; three fractions will be administered
  Other Names: Steretactic body radiotherapy

SUMMARY:
Aim of this study is to evaluate if low-dose radiotherapy (LDR) can intensify local effect of a chemotherapy regimen with Gem-based doublets administered sequentially with stereotactic body radiotherapy (SBRT) and to assess the safety and efficacy of this combined treatment on patients affected by locally advanced pancreatic adenocarcinoma (LAPC).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of the pancreas
* Patients with unresectable disease based on institutional standardized criteria of unresectability or patients whose disease appeared potentially resectable on axial CT imaging but were found unresectable at surgery
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2. Age ≥ 18
* Patients with biliary or gastroduodenal obstruction must have drainage or surgical bypass prior to starting treatment
* Patients with radiographically assessable disease
* Adequate bone marrow, hepatic and renal function: -Hemoglobin >10.0 g/dL, absolute neutrophil count > 1.5 x 10^9/L, platelet count > 100 x 10^9/L. -Aspartate transaminase (AST or SGOT) and alanine transaminase (ALT or SGPT) should be ≤ 3 x upper limit of normal (ULN). -Total bilirubin < 2 mg/dL. Patients with elevated bilirubin due to obstruction should be stented and their bilirubin should decrease to < 2 mg/dL prior to study entry. - Creatinine < 3 mg/dL or Creatinine clearance > 40 mL/min (calculated according to Cockroft and Gault)

Exclusion Criteria:

* Evidence of metastatic disease in the major viscera or peritoneal seeding or ascites
* Gastric or duodenal obstruction
* Previous peripheral neuropathy
* Previous irradiation to the planned field; previous chemotherapy for pancreatic cancer
* Malignancy (within the past two years) except non-melanomatous skin cancer or carcinoma in situ of the cervix, uterus, or bladder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2014-01; Primary Completion 2023-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 1 year
  defined as the time from the initiation of therapy to the time of first event (local, regional or distant progression or death due to any cause). Patients without any such event at the time of data analysis will be censored at the last date they were known to be event-free. Patients with no tumor assessments after baseline will be censored at day 1

SECONDARY OUTCOMES:
Toxicity(scored according to the National Cancer Institute Common Terminology Criteria for Adverse Events (v4.0)) | every 3 months, up to 1 year
  Acute gastrointestinal toxicity is defined as adverse events occurring <3 months after SBRT; long-term toxicity was defined as those occurring after 3 months. Toxicity is scored according to the National Cancer Institute Common Terminology Criteria for Adverse Events (v4.0)
Overall survival | 1 year
  defined as the time from the date of initiation of therapy to date of death due to any cause. Patients who is alive on the date of last follow-up were censored on that date

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Meduri, MD, Principal Investigator — Azienda Ospedaliero-Universitaria Policlinico di Modena
Locations (1):
- Azienda Ospedaliero-Universitaria Policlinico di Modena, Modena, MO, Italy

REFERENCES:
- [Background] Mantini G, Valentini V, Meduri B, Margaritora S, Balducci M, Micciche F, Nardone L, De Rose F, Cesario A, Larici AR, Maggi F, Calcagni ML, Granone P. Low-dose radiotherapy as a chemo-potentiator of a chemotherapy regimen with pemetrexed for recurrent non-small-cell lung cancer: a prospective phase II study. Radiother Oncol. 2012 Nov;105(2):161-6. doi: 10.1016/j.radonc.2012.09.006. Epub 2012 Oct 12. PMID 23068709
- [Background] Regine WF, Hanna N, Garofalo MC, Doyle A, Arnold S, Kataria R, Sims J, Tan M, Mohiuddin M. Low-dose radiotherapy as a chemopotentiator of gemcitabine in tumors of the pancreas or small bowel: a phase I study exploring a new treatment paradigm. Int J Radiat Oncol Biol Phys. 2007 May 1;68(1):172-7. doi: 10.1016/j.ijrobp.2006.11.045. Epub 2007 Feb 2. PMID 17276612
- [Background] Mahadevan A, Jain S, Goldstein M, Miksad R, Pleskow D, Sawhney M, Brennan D, Callery M, Vollmer C. Stereotactic body radiotherapy and gemcitabine for locally advanced pancreatic cancer. Int J Radiat Oncol Biol Phys. 2010 Nov 1;78(3):735-42. doi: 10.1016/j.ijrobp.2009.08.046. Epub 2010 Feb 18. PMID 20171803
- [Background] Valentini V, Massaccesi M, Balducci M, Mantini G, Micciche F, Mattiucci GC, Dinapoli N, Meduri B, D'Agostino GR, Salvi G, Nardone L. Low-dose hyperradiosensitivity: is there a place for future investigation in clinical settings? Int J Radiat Oncol Biol Phys. 2010 Feb 1;76(2):535-9. doi: 10.1016/j.ijrobp.2009.02.075. Epub 2009 Jun 18. PMID 19540061